CLINICAL TRIAL: NCT04356833
Title: A Pilot, Open Label, Phase II Clinical Trial of Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA)
Brief Title: Nebulised Rt-PA for ARDS Due to COVID-19
Acronym: PACA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 132151
Record Dates: First submitted 2020-04-14; First posted 2020-04-22 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: COVID

STUDY DESIGN:
Intervention Model Description: phase II, open label, uncontrolled, repeated dose, pilot trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Nebulised recombinant tissue-Plasminogen Activator (rt-PA) - cohort 1 (Experimental): Patients in the rt-PA group received the first dose as soon as possible after registration.
  Initial dosing regime: 10 mg of rt-PA dissolved in 5 ml of diluent given every 6 hrs (resulting in a total daily dose of 40mg) for a maximum of 66 hrs, in addition to standard of care for COVID-19 acute respiratory distress syndrome (ARDS). Following protocol amendment, dosing duration was increased from 3 days to up to 14 days of rt-PA treatment. Six patients were receiving Invasive mechanical ventilation and 3 were receiving non-invasive ventilation.
  Interventions: Drug: Nebulised recombinant tissue-Plasminogen Activator (rt-PA) - Cohort 1
- Historical matched controls - cohort 1 (No Intervention): Historical matched controls were recruited at a ratio of 2 controls to every 1 rtPA + SOC arm patient, and were matched according to the following characteristics:
  1. Ventilation and oxygen type (IMV and non-invasive oxygen support)
  2. Severity as determined by PaO2/FiO2 ratio
  3. Gender
  4. Age (+/- 2 years, up to a maximum of 10 years)
  5. Ethnicity
- Nebulised recombinant tissue-Plasminogen Activator (rt-PA) - cohort 2 IMV (Experimental): In cohort 2, fewer timepoints were collected, which allowed for more rapid recruitment while at the same time not compromising safety monitoring. A more flexible dosing regimen for rtPA was utilised.
  Patients on IMV received 60mg daily over three doses for up to 14 days
  Interventions: Drug: Nebulised recombinant tissue-Plasminogen Activator (rt-PA) - Cohort 2 IMV
- Nebulised recombinant tissue-Plasminogen Activator (rt-PA) - cohort 2 NIV (Experimental): n cohort 2, fewer timepoints were collected, which allowed for more rapid recruitment while at the same time not compromising safety monitoring. A more flexible dosing regimen for rtPA was utilised.
  Patients on NIV received 60mg daily for over 3 doses for two days, followed by 12 days receiving 40mg daily over two doses.
  Interventions: Drug: Nebulised recombinant tissue-Plasminogen Activator (rt-PA) - Cohort 2 NIV

INTERVENTIONS:
Drug: Nebulised recombinant tissue-Plasminogen Activator (rt-PA) - Cohort 1 — Patients in the rt-PA group received the first dose as soon as possible after registration.
  Initial dosing regime: 10 mg of rt-PA dissolved in 5 ml of diluent given every 6 hrs (resulting in a total daily dose of 40mg) for a maximum of 66 hrs, in addition to standard of care for COVID-19 acute respiratory distress syndrome (ARDS). Following protocol amendment, dosing duration was increased from 3 days to up to 14 days of rt-PA treatment.
  Other Names: Cohort 1
  Arms: Nebulised recombinant tissue-Plasminogen Activator (rt-PA) - cohort 1
Drug: Nebulised recombinant tissue-Plasminogen Activator (rt-PA) - Cohort 2 IMV — Patients on IMV received 60mg daily over three doses for up to 14 days
  Other Names: Cohort 2 IMV
  Arms: Nebulised recombinant tissue-Plasminogen Activator (rt-PA) - cohort 2 IMV
Drug: Nebulised recombinant tissue-Plasminogen Activator (rt-PA) - Cohort 2 NIV — NIV patients received 60mg daily over 3 doses for two days, followed by 12 days receiving 40mg daily over two doses.
  Other Names: Cohort 2 NIV
  Arms: Nebulised recombinant tissue-Plasminogen Activator (rt-PA) - cohort 2 NIV

SUMMARY:
Some patients infected with COVID-19 develop a severe form of a lung disease called acute respiratory distress syndrome (ARDS). In these patients, the lungs become severely inflamed because of the virus. The inflammation causes fluid from nearby blood vessels to leak into the tiny air sacs in the lungs, making breathing increasingly difficult. This fluid forms small clots in the air sacs. In some patients, these clots do not disappear in a timely fashion. Furthermore, the small clots in the air sacs obstruct the air and oxygen getting deep into the lungs, interfering with ventilation. The trial recruited patients with COVID-19 induced ARDS. Eligible patients (or if patients lack capacity, their legal representative) were provided with an information sheet and informed consent was sought. Eligibility was mainly assessed via routine clinical assessments. Patients received a nebulised version of a type of drug called tissue plasminogen activator (rt-PA) that was inhaled using a nebuliser. This is normally a drug used to break down blood clots. In the nebulised form, we hypothesised that it may be useful for stopping clots forming in the lungs. The study ran two cohorts sequentially. In cohort 1, 9 consented patients received nebulised rtPA in addition to SOC. As an observational arm, matched historical controls who received SOC were also recruited at a ratio of 2 controls to every 1 treatment arm patient, resulting in 18 historical controls. After the first wave of COVID-19 cases decreased in August 2020 in the UK, it became difficult to continue recruiting, so recruitment was closed for cohort 1. With a second surge in early 2021, cohort 2 opened with the aim to recruit more patients to provide more data on the safety of rt-PA. In cohort 2, fewer timepoints were collected, which allowed for more rapid recruitment without compromising safety monitoring. A more flexible dosing regimen for rtPA was utilised. 26 patients were recruited in total, 12 in the IMV arm and 14 in the NIV/NIRS arm. To evaluate drug efficacy, the improvement of oxygen levels over time and safety were monitored throughout. Blood samples were taken to measure markers of clotting and inflammation in both cohorts. From the end of the treatment phase, both groups were followed up in accordance with SOC up to a maximum of 28 days, starting from the day of first dose of rt-PA.

DETAILED DESCRIPTION:
This is a phase II, open label, uncontrolled, repeated dose, pilot trial of nebulised rt-PA in patients with COVID-19 ARDS.

The study recruited patients requiring either invasive mechanical ventilation (IMV) or non-invasive ventilation/non-invasive respiratory support (NIV/NIRS) between April 2020 and February 2021. Eligible patients (or if patients lacked capacity, their legal representative) were provided with an information sheet and informed consent was sought. Eligibility was assessed via routine clinical assessments, which may have been done prior to consent. The only exceptions were pregnancy tests (blood or urine), and possibly any assessments that were not done as per routine care. If required, these would have been done following consent, and all screening assessments must have been done during the 24-hour period before dosing with rt-PA.

In the rt-PA treatment group of cohort 1, 9 consented patients received nebulised rt-PA in addition to standard of care (SOC). Out of the 9 patients, 6 were on the IMV arm and another 3 were on the NIV arm. As an observational arm, matched historical controls who received only SOC were also recruited at a ratio of 2 controls to every 1 treatment arm patient, to ensure that any changes were not entirely due to disease resolution. A total of 18 patients were recruited to the historical matched control arm of cohort 1. Therefore a total of 27 patient constituted cohort 1.

For patients in the treatment group, 10 mg of rt-PA dissolved in 5 ml of diluent was given every 6 hrs for 3 days. This was extended to up to 14 days with a subsequent protocol amendment. Dose modifications were not permitted. Efficacy was described as the change in PaO2/FiO2 ratio from baseline, daily during treatment, end of treatment, 3 days post end of treatment and 5 days post end of treatment.

With a second surge of COVID-19 in early 2021, cohort 2 was opened to recruit more patients to provide additional data on the safety of rt-PA. Fewer timepoints were collected, which allowed for more rapid recruitment while at the same time not compromising safety monitoring. A more flexible dosing regimen for rt-PA was utilised. Patients on IMV received 60mg daily over three doses for up to 14 days. NIV patients received 60mg daily over 3 doses for two days, followed by 40mg daily over two doses for up to 12 days. A total of 26 patients were recruited in cohort 2, 12 on the IMV arm and 14 on the NIV/NIRS arm.

From the end of the treatment phase (after Day 14), patients were followed up in accordance with SOC for 28 days from the day of first dose of rtPA.

Safety monitoring was performed by assessment of the incidence and severity of bleeding events, and by the monitoring of plasma fibrinogen levels and routine coagulation parameters. Additional samples were taken for exploratory assessment of potential biomarkers, including, but not restricted to, PAI- 1, alpha 2 antiplasmin and a range of inflammatory cytokines and coagulation proteins. All other monitoring was done as per SOC.

A Data Monitoring Committee (DMC) was set-up to review safety data within the trial along with the final study results and advise on progressing from a pilot study to a randomised control trial based on the safety and efficacy data that was to be collected. If a patient had major pulmonary bleeding at any time, further dosing of patients was to be stopped and an ad-hoc DMC review to be arranged before resuming dosing (see section 12.2 Data Monitoring Committee).

Although there is extensive experience with the use of nebulised rt-PA in the context of the underlying inflammation, safety measures were included in the study. A gap of 24hrs was maintained between the first and second patient. At 24hrs, if patient 1 had no evidence of major pulmonary bleeding suggesting exaggerated alveolar fibrinolysis and no evidence of fibrinogen reduction of more than 50% (suggestive of systemic absorption), then the second patient was to be dosed. Both patients were evaluated for 72 hrs post dose for any major pulmonary bleeding and if no bleeding was noticed, then the rest of the cohort were to be recruited after the review of the safety data by the trial management group comprised of the investigators. Any concerns with the data were referred to the DMC for review. If the safety profile was acceptable, dosing of the third and subsequent patients in the rt-PA group would resume with no required interval between patients.

A statistically powered randomised controlled trial (RCT) would be ideal to define the magnitude of benefit and impact on overall survival and is the typical design in patients with ARDS. Although there is clinical data on the safety of nebulised rt-PA, there is no data in this clinical condition to facilitate a sample size calculation. There is data from a small RCT that has used another fibrinolytic agent, but the doses were not comparable. When a patient is randomised to receive no treatment, this precludes participation in other interventional studies which might decrease the risk of mortality. The most recent figures suggest a 50% mortality in patients receiving IMV. Currently there is a concerted effort to introduce multiple therapies based on our understanding of the pathophysiologic basis of the disorder. Further, if this pilot study shows significant effect in a subset of patients, there would be justification to progress to a statistically powered RCT. In the event of major adverse drug reactions or minor improvement in the oxygenation as assessed by PaO2/FiO2 , there are minimal gains to be had with a larger randomised control study.

ELIGIBILITY:
Inclusion Criteria (cohorts 1 and 2):

1. Patients with COVID-19 (confirmed by PCR or radiologically)
2. ≥16 years
3. Willing and able to provide written informed consent or where patient doesn't have capacity, consent obtained from a legal representative
4. Patients on IMV must meet both the following criteria:

   1. PaO2/FiO2 of ≤ 300 (definition of ARDS)
   2. Intubated > 6 hrs
5. Patients not intubated must meet the following criteria:

   1. PaO2/FiO2 ≤ 300 or equivalent imputed by non-linear calculation from SpO2/FiO2 (see look-up table in appendices)
   2. In-patient >6 hours and being actively treated
   3. On support with non-invasive ventilation OR continuous positive airway pressure (CPAP) OR high flow OR standard oxygen therapy

Exclusion Criteria (cohort 1):

1. Females who are pregnant
2. Concurrent involvement in another experimental investigational medicinal product
3. Known allergies to the IMP or excipients of IMP
4. A pre-existing bleeding disorder (e.g. severe haemophilia) with no definitive treatment
5. Pre-existing severe cardiopulmonary disease (e.g. incurable lung cancer, severe chronic obstructive lung disease, cardiomyopathy, heart failure or impaired contractility <estimated 40% LVEF or RVEF)
6. Fibrinogen < 2.0 g/L at time of screening
7. Patients considered inappropriate for active treatment (e.g. being considered for palliative care)
8. Patients with active bleeding in the preceding 7 days
9. Patients who in the opinion of the investigator are not suitable

Exclusion Criteria (cohort 2):

1. Females who are pregnant
2. Known allergies to the IMP or excipients of IMP
3. Fibrinogen < 1.5 g/L at time of screening
4. Patients considered inappropriate for active treatment (e.g. being considered for palliative care)
5. Patients who in the opinion of the investigator are not suitable

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pratima Chowdary, Principal Investigator — Royal Free London NHS Foundation Trust
Locations (1):
- The Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Cohort 1, as an observational arm, matched historical controls who received SOC were also recruited at a ratio of 2 controls to every 1 treatment arm patient, resulting in 18 historical controls.
Groups:
- Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1: nebulised recombinant tissue-Plasminogen Activator (rt-PA) - Cohort 1: Patients in the cohort 1 rt-PA group received the first dose as soon as possible after registration.
- Historical Matched Controls - Cohort 1: Matched historical controls who received standard of care were recruited at a ratio of 2 controls to every 1 treatment arm.
- Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV Arm: nebulised recombinant tissue-Plasminogen Activator (rt-PA) - cohort 2 IMV arm - Patients on IMV received 60mg daily over three doses for up to 14 day
- Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV Arm: nebulised recombinant tissue-Plasminogen Activator (rt-PA) - cohort 2 NIV arm -NIV patients received 60mg daily over 3 doses for two days, followed by 12 days receiving 40mg daily over two doses (for a maximum of 12 days, and doses were changed if patient required IMV)
Period: Overall Study
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Historical Matched Controls - Cohort 1 | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV Arm | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV Arm
Started | 9 | 18 | 12 | 14
Completed | 9 | 18 | 12 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis of C1 and C2 was undertaken separately.
Groups:
- Historical Matched Controls - Cohort 1: Matched historical controls who received standard of care were also recruited at a ratio of 2 controls to every 1 treatment arm patient. Matching was done according to the following criteria in the order stated:
  1. Ventilation and oxygen type (IMV and non-invasive oxygen support)
  2. Severity as determined by PaO2/FiO2 ratio
  3. Gender
  4. Age (+/- 2 years, up to a maximum of 10 years)
  5. Ethnicity
- Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV: In cohort 2, fewer timepoints were collected, which allowed for more rapid recruitment while at the same time not compromising safety monitoring. A more flexible dosing regimen for rtPA was utilised.
  Patients on NIV received 60mg daily for over 3 doses for two days, followed by 12 days receiving 40mg daily over two doses (for a maximum of 12 days, and doses were changed if patient required IMV).
- Total: Total of all reporting groups
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Historical Matched Controls - Cohort 1 | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV | Total
Number analyzed (Participants) | 9 | 18 | 12 | 14 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 8 | 8 | 8 | 28
  >=65 years | 5 | 10 | 4 | 6 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 5 | 2 | 21
  Male | 4 | 9 | 7 | 12 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 14 | 12 | 11 | 46
  Unknown or Not Reported | 0 | 4 | 0 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 3 | 6 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 6 | 10 | 4 | 4 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 5 | 3 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 9 | 18 | 12 | 14 | 53
PaO2/FiO2 Ratio [Mean (Standard Deviation); unit: mmHg (rounded)] — Cohort 1: All available P/F ratio values were extracted per day and summarised every 4 hours (± 2h). Time 0 is baseline. Cohort 2: Up to six P/F ratio values were extracted per day including the worst P/F ratio over the preceding one day; however, the analysis for Cohort 2 includes only the lowest value for the day.
  mmHg (rounded) | 154 (53) | 154 (73) | 120 (28) | 126 (42) | 139 (55)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy - PaO2/FiO2 Ratio
Description: PaO2/FiO2 measured at multiple timepoints: baseline, during treatment, end of treatment, 3 days post end of treatment and 5 days post end of treatment. For Cohort 1, all available values were extracted per day and summarised every 4 hours (± 2h). For Cohort 2, up to six values were extracted per days including the worst ratio over the preceding day; Cohort 2 included only the lowest value for the day. PaO2/FiO2 ratio is the ratio of arterial oxygen partial pressure to fractional inspired oxygen. It is a widely used clinical indicator of hypoxaemia and is used to classify severity of acute respiratory distress syndrome. Limited data was observed due to patient discharge or death: Day 14 is presented below, and the last value available on treatment regardless of the duration of treatment (death or discharge may have occurred within 14 days) was summarised post-hoc. Summarized values were rounded to the nearest integer.
Time Frame: Day 14 and last value available on treatment (which could occur up to 14 days, death or discharge may have occurred within 14 days)
Population: Limited data was observed due to patient discharge or death: Day 14 is presented below, and the last value available on nebulized Rt-PA treatment regardless of the duration of nebulized Rt-PA treatment (death or discharge may have occurred within 14 days) was summarised post-hoc. The historical matched controls were not treated with nebulized Rt-PA and therefore no data is available in the post-hoc analysis of the last on-treatment day.
Measure: Mean (Standard Deviation); unit: mmHg (rounded)
Groups:
- Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV: Nebulised recombinant tissue-Plasminogen Activator (rt-PA) - Cohort 2 invasive mechanical ventilation
- Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV: Nebulised recombinant tissue-Plasminogen Activator (rt-PA) - Cohort 2 non-invasive ventilation/non-invasive respiratory support
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Historical Matched Controls - Cohort 1 | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV
Number analyzed (Participants) | 9 | 4 | 12 | 14
mmHg (rounded)
  Day 14: number analyzed (Participants) | 2 | 4 | 8 | 5
  Day 14 | 227 (83) | 209 (49) | 155 (104) | 248 (89)
  Last On-Treatment Day: number analyzed (Participants) | 9 | 0 | 12 | 14
  Last On-Treatment Day | 218 (73) |  | 169 (108) | 240 (104)

2. Primary Outcome: Safety- Participants With Major Bleeding Events Directly Attributable to Study Drug
Description: Number of patients with major bleeding events assessed as related to the study drug summarised in each group.
Time Frame: 28 days
Population: Bleeding events were not recorded in historical matched controls (cohort 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV
Number analyzed (Participants) | 9 | 12 | 14
Participants | 0 | 1 | 0

3. Primary Outcome: Safety- Participants With Serious Adverse Events Causally Related to Treatment
Description: Number of Participants with serious adverse events causally related to treatment.
  Adverse events (other than bleeding events) were not recorded in the study.
Time Frame: 28 days
Population: Bleeding events were not recorded in historical matched controls (cohort 1) Adverse events (other than bleeding events) were not recorded in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV
Number analyzed (Participants) | 9 | 12 | 14
Participants | 0 | 0 | 0

4. Primary Outcome: Safety- Participants With Decrease in Fibrinogen Levels to < 1gm/L
Description: Number of participants with a decrease in fibrinogen levels to < 1gm/L during the treatment period and 48 hours after the last dose.
Time Frame: 28 days
Population: Fibrinogen levels were not recorded for the historical matched controls (cohort 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV
Number analyzed (Participants) | 9 | 12 | 14
Participants | 0 | 0 | 0

5. Secondary Outcome: Lung Compliance
Description: Changes in lung compliance (defined as tidal volume / (peak inspiratory pressure - PEEP) from baseline (same day as start of treatment but prior to start of treatment) was a secondary outcome as defined in the protocol. Limited data was observed due to patient discharge or death, therefore the last value available on treatment regardless of the duration of treatment (death or discharge may have occurred within 14 days) was summarised post-hoc and presented below. For cohort 2, the daily measurement coinciding with the worst PF ratio (as close as possible in date and time) was used for the summaries.
Time Frame: Last value available on treatment (which could occur up to 14 days, death or discharge may have occurred within 14 days)
Population: Lung compliance was not recorded in the historical matched controls (cohort 1) or in patients in the NIV group. During the COVID pandemic, investigations and observations were done less rigorously than compared to routine care. Many of the secondary outcome measures were based on the standard of care rather than being study specific observations.
Measure: Mean (Standard Deviation); unit: mL/cmH2O
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV
Number analyzed (Participants) | 6 | 12
mL/cmH2O | 40.4 (22.5) | 37.6 (42.8)

6. Secondary Outcome: Clinical Status as Determined by a 7-point WHO Ordinal Scale
Description: Clinical status as assessed by a 7-point WHO ordinal scale at baseline and daily up to 5 days post end of treatment and at day 28, discharge or death (whichever comes first).
  1. Limitation of activities
  2. Hospitalized, no oxygen therapy
  3. Oxygen by mask or nasal prongs
  4. Non-invasive ventilation or high-flow oxygen
  5. Intubation and mechanical ventilation
  6. Ventilation+ additional organ support (vasopressor, RRT, ECMO)
  7. Death
Time Frame: Day 28
Population: This outcome measure was modified between cohort 1 and 2, and the 7-point WHO scale was only collected from patients in cohort 2. Limited data was observed due to patient discharge or death, therefore only data for cohort 2 are presented. During the COVID pandemic, investigations and observations were done less rigorously than compared to routine care. Many of the secondary outcome measures were based on the standard of care rather than being study specific observations.
Measure: Count of Participants; unit: Participants
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV
Number analyzed (Participants) | 12 | 14
Participants
  1. Limitation of activities | 0 | 0
  2. Hospitalized, no oxygen therapy | 0 | 0
  3. Oxygen by mask or nasal prongs | 1 | 2
  4. Non-invasive ventilation or high-flow oxygen | 0 | 0
  5. Intubation and mechanical ventilation | 2 | 0
  6. Ventilation+ additional organ support vasopressor, RRT, ECMO) | 1 | 0
  7. Death | 0 | 0
  Data Missing | 8 | 12

7. Secondary Outcome: Sequential Organ Failure Assessment (SOFA) Score
Description: The Sequential Organ Failure Assessment (SOFA) is a morbidity severity score and mortality estimation tool developed from a large sample of ICU patients throughout the world. The SOFA was designed to focus on organ dysfunction and morbidity, with less of an emphasis on mortality prediction. It requires the following (worst value within past 24 hours): FiO2, PaO2, Mechanical ventilation, Platelets, Bilirubin, Glasgow coma scale, Mean arterial pressure, Vasopressors, Creatinine, Urine output, and can be calculated by entering the results above into an online tool: https://clincalc.com/IcuMortality/SOFA.aspx. The SOFA Score is a mortality prediction score that is based on the degree of dysfunction of six organ systems. A higher value for each organ system is associated with higher mortality, and here total score was used. The total possible score ranges from 0 to 24.
Time Frame: 28 days (day 14 presented)
Population: During the COVID pandemic, investigations and observations were done less rigorously than compared to routine care. Many of the secondary outcome measures were based on the standard of care rather than being study specific observations.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV: INebulised recombinant tissue-Plasminogen Activator (rt-PA) - Cohort 2 invasive mechanical ventilation
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Historical Matched Controls - Cohort 1 | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV
Number analyzed (Participants) | 7 | 2 | 6 | 4
score on a scale | 7.71 (4.82) | 7 (7.07) | 10.7 (1.63) | 4.8 (4.92)

8. Secondary Outcome: Number of Oxygenation Free Days
Description: Number of oxygen free days, up to 28 days or death or discharge, whichever occured first.
Time Frame: up to 28 days or death or discharge, whichever occurred first
Measure: Median (Full Range); unit: days
Groups:
- Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1: Nebulised recombinant tissue-Plasminogen Activator (rt-PA) - Cohort 1
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Historical Matched Controls - Cohort 1
Number analyzed (Participants) | 12 | 14 | 9 | 18
days | 0 [0 to 5] | 0.5 [0 to 6] | 0 [0 to 10] | 0 [0 to 12]

9. Secondary Outcome: Number of Ventilator Free Days
Description: Number of ventilator free days, up to 28 days or death or discharge, whichever occured first
Time Frame: up to 28 days or death or discharge, whichever occured first
Measure: Median (Full Range); unit: Days
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Historical Matched Controls - Cohort 1
Number analyzed (Participants) | 12 | 14 | 6 | 10
Days | 0 [0 to 8] | 7.5 [0 to 23] | 0 [0 to 13] | 1.5 [0 to 13]

10. Secondary Outcome: Intensive Care Stay
Description: Intensive care stay, up to 28 days or death or discharge, whichever occurs first, was a secondary outcome as defined in the protocol. However, due to protocol amendments, difficulties in collecting this data, differences in study design between cohort 1 and cohort 2 and limited comparability of this outcome measure between groups, results are presented but have limited interpretation and should not be used or compared. For cohort 1, the number of days in ICU were limited to the 1st admission.
Time Frame: 28 days
Population: Due to protocol amendments, difficulties in collecting this data (owing to a combination of death, recovery and a smaller data set used for monitoring patients during COVID), differences in study design between cohort 1 & cohort 2, and limited comparability of this outcome measure between groups, results are presented but have limited interpretation and should not be used or compared. For cohort 1, the number of days in ICU were limited to the 1st admission.
Measure: Median (Full Range); unit: Days
Groups:
- Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV Arm: nebulised recombinant tissue-Plasminogen Activator (rt-PA) - cohort 2 NIV arm -NIV patients received 60mg daily over 3 doses for two days, followed by 12 days receiving 40mg daily over two doses.
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Historical Matched Controls - Cohort 1 | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV Arm | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV Arm
Number analyzed (Participants) | 8 | 12 | 8 | 2
Days | 19 [5 to 28] | 12 [2 to 28] | 9 [1 to 13] | 5 [1 to 8]

11. Secondary Outcome: Number of Days of New Mechanical Ventilation Use During in the First 28 Days
Description: incidence and number of days of new mechanical ventilation use during in the first 28 days was a secondary outcome measure as defined in the protocol.
Time Frame: 28 days
Measure: Median (Full Range); unit: Days
Groups:
- Historical Matched Controls - Cohort 1: Matched historical controls who received standard of care were recruited at a ratio of 2 controls to every 1 treatment arm in cohort 1.
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Historical Matched Controls - Cohort 1
Number analyzed (Participants) | 12 | 14 | 6 | 10
Days | 14.5 [2 to 23] | 0 [0 to 12] | 23 [13 to 28] | 10.5 [2 to 28]

12. Secondary Outcome: Number of Days of Non-invasive Ventilation Use
Description: Number of days of new oxygen use, non-invasive ventilation or high flow oxygen devices
Time Frame: Day 28
Measure: Median (Full Range); unit: days
Groups:
- Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 NIV: Nebulised recombinant tissue-Plasminogen Activator (rt-PA) - Cohort 1 non-invasive ventilation/non-invasive respiratory support
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 NIV | Historical Matched Controls - Cohort 1
Number analyzed (Participants) | 12 | 14 | 2 | 5
days | 0.5 [0 to 8] | 6 [0 to 23] | 6.5 [5 to 8] | 3 [1 to 3]

13. Secondary Outcome: In-hospital Mortality
Description: In-hospital mortality.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Historical Matched Controls - Cohort 1 | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV
Number analyzed (Participants) | 9 | 18 | 12 | 14
Participants | 1 | 10 | 5 | 3

14. Post Hoc Outcome: Number of Ventilator Free Days (With Imputation)
Description: Number of ventilator free days, up to 28 days or death or discharge, whichever occurs first was a secondary outcome as defined in the protocol. However, a post-hoc exploration of the data recalculated the number of ventilator free days, taking into account the number of days post-discharge. For this new calculation, days post-discharge up to 28 days, were assumed to be days when the patient did not receive oxygen or ventilation.
  .
Time Frame: up to 28 days or death, whichever occurred first
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV | Historical Matched Controls - Cohort 1
Number analyzed (Participants) | 6 | 12 | 14 | 10
days | 4.3 (6.8) | 5.75 (9.94) | 21.4 (9.68) | 8.4 (9.6)

15. Post Hoc Outcome: Number of Oxygen Free Days (With Imputation)
Description: Number of oxygen free days, up to 28 days or death or discharge, whichever occurs first was a secondary outcome as defined in the protocol. However, a post-hoc exploration of the data recalculated the number of Oxygen free days, taking into account the number of days post-discharge. For this new calculation, days post-discharge up to 28 days, were assumed to be days when the patient did not receive oxygen or ventilation.
Time Frame: up to 28 days or death, whichever occurred first
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV | Historical Matched Controls - Cohort 1
Number analyzed (Participants) | 9 | 12 | 14 | 18
days | 6.2 (9.5) | 4.42 (8.1) | 13.43 (11.1) | 6.7 (9.2)

16. Post Hoc Outcome: Number of Particpants With "New IMV (Deterioration)"
Description: Incidence and number of days of new mechanical ventilation use during in the first 28 days was a secondary outcome measure as defined in the protocol. However, a post-hoc exploration of the data redefined "New IMV (deterioration)" as any patient requiring mechanical ventilation (IMV) after a period of non-mechanical ventilation after receiving r-tPA.
Time Frame: 28 days
Population: New IMV (deterioration) was not recorded in the historical matched controls (cohort 1). During the COVID pandemic, investigations and observations were done less rigorously than compared to routine care. Many of the secondary outcome measures were based on the standard of care rather than being study specific observations.
Measure: Count of Participants; unit: Participants
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV
Number analyzed (Participants) | 9 | 12 | 14
Participants | 0 | 1 | 2

17. Post Hoc Outcome: Numer of Participants With "New Oxygen Use (Relapse)"
Description: Incidence and number of days of new oxygen use, non-invasive ventilation or high flow oxygen devices in the first 28 days was a secondary outcome as defined in the protocol, however a post-hoc clarification of the endpoint redefined "New Oxygen use (relapse)" as any patient requiring oxygen support after being on room air for a whole day.
Time Frame: 28 days
Population: New oxygen use was not recorded in the historical matched controls (cohort 1). During the COVID pandemic, investigations and observations were done less rigorously than compared to routine care. Many of the secondary outcome measures were based on the standard of care rather than being study specific observations.
Measure: Count of Participants; unit: Participants
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV
Number analyzed (Participants) | 9 | 12 | 14
Participants | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Maximum of 28 days per patient, starting from dosing day 1
Description: Only serious adverse events related to the IMP, and all bleeding events were collected/reported. Bleeding events were identified as adverse events of special interest (AESI). In addition, the ISTH (International Society of Haemostasis and Thrombosis) classification for bleed severity as used for anticoagulation studies was implemented.
  Events were not collected/recorded in historical matched controls (cohort 1).
Groups:
- Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1: Patients in the rt-PA group received the first dose as soon as possible after registration.
  Initial dosing regime: 10 mg of rt-PA dissolved in 5 ml of diluent given every 6 hrs (resulting in a total daily dose of 40mg) for a maximum of 66 hrs, in addition to standard of care for COVID-19 acute respiratory distress syndrome (ARDS).
  Following a protocol amendment, dosing duration was increased from 3 days to up to 14 days of rt-PA treatment. Six patients were receiving Invasive mechanical ventilation and 3 were receiving non-invasive ventilation.
- Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV: In cohort 2, fewer timepoints were collected, which will allowed for more rapid recruitment while at the same time not compromising safety monitoring. A more flexible dosing regimen for rtPA was utilised.
  Patients on IMV received 60mg daily over three doses for up to 14 days
- Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV: In cohort 2, fewer timepoints were collected, which will allowed for more rapid recruitment while at the same time not compromising safety monitoring. A more flexible dosing regimen for rtPA was utilised.
  Patients on NIV received 60mg daily for over 3 doses for two days, followed by 12 days receiving 40mg daily over two doses.
Arm/Group | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 | Historical Matched Controls - Cohort 1 | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV
All-Cause Mortality (participants affected / at risk) | 1/9 | 10/18 | 5/12 | 3/14
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/0 | 1/12 | 0/14
Other Adverse Events (participants affected / at risk) | 4/9 | 0/0 | 9/12 | 4/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 (N=9) | Historical Matched Controls - Cohort 1 (N=0) | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV (N=12) | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV (N=14)
Cerebral bleed (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Events were not collected/recorded in historical matched controls (cohort 1).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 1 (N=9) | Historical Matched Controls - Cohort 1 (N=0) | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 IMV (N=12) | Nebulised Recombinant Tissue-Plasminogen Activator (Rt-PA) - Cohort 2 NIV (N=14)
Bleed: Central venous catheters access site (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Events were not collected/recorded in historical matched controls (cohort 1).
Gastro-intestinal bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) — Events were not collected/recorded in historical matched controls (cohort 1).
Blood-stained tracheobronchial secretion (Surgical and medical procedures) | 1 (1) | 0 (0) | 7 (12) | 1 (2) — Events were not collected/recorded in historical matched controls (cohort 1).
Tracheostomy site bleed (Surgical and medical procedures) | 2 (2) | 0 (0) | 1 (1) | 0 (0) — Events were not collected/recorded in historical matched controls (cohort 1).
Bleed: chest-drain related (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Events were not collected/recorded in historical matched controls (cohort 1).
Epistaxis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) — Events were not collected/recorded in historical matched controls (cohort 1).
Other (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) — Events were not collected/recorded in historical matched controls (cohort 1).

LIMITATIONS AND CAVEATS:
Open label design with a small sample size, missing data and absence of a concurrent control group. A change in a patient's condition could result in an alteration in ventilation type post-enrolment, or in discharge. Furthermore, the P/F ratio was calculated by different methods: for those receiving NIRS, the P/F ratio was determined by converting SpO2 and oxygen flow rate, whereas the P/F ratio was readily available for IMV group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT04356833/Prot_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan - cohort 2 (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT04356833/SAP_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan - cohort 1 (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT04356833/SAP_002.pdf